CLINICAL TRIAL: NCT01086514
Title: Dual Energy Contrast Enhanced Digital Mammography for the Detection and Preoperative Staging of Breast Cancer
Brief Title: Digital Mammography for the Detection and Preoperative Staging of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-024
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Breast; mammography; MRI; Digital Mammography; 10-024
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Dual Energy Contrast Enhanced Digital Mammography (DE CEDM) (Experimental): In this study we will perform Dual Energy Contrast Enhanced Digital Mammography (DE CEDM) on patients with newly diagnosed breast cancer using a dedicated research system, derived from a standard digital mammography unit and review workstation (Senographe DS and SenoAdvantage) modified to deliver the required dual energy paired exposures and visualization of combined images.
  Interventions: Procedure: Dual Energy Contrast Enhanced Digital Mammography (DE CEDM)

INTERVENTIONS:
Procedure: Dual Energy Contrast Enhanced Digital Mammography (DE CEDM) — Each patient will have: Bilateral digital mammography, Bilateral Breast MRI, Bilateral Contrast Enhanced Digital Mammography. The latter examination is the only change in patient management. An additional contrast injection is involved. Results of the DE CEDM will be compared with routine digital mammography and breast MRI. The reference standard is pathology. If surgery is to be done; every attempt will be made to perform all imaging exams within 30 days.

SUMMARY:
Breast tumors are normally seen with mammography or ultrasound without the use of a dye but the size and extent of the tumor may be hard to see. Currently, after initial mammography, many patients undergo bilateral breast MR to further stage the local tumor. It is able to not only detect anatomic abnormalities but can also evaluate changes such as the development of new blood vessels, which occurs with the development of cancers. MRI is extremely sensitive and detects unsuspected disease in up to 25% of patients, which affects their treatment. It also detects unsuspected cancer in the other breast in some patients.

However, MRI is expensive, not always available, and some patients are unable to undergo MRI due to the presence of pacemakers, clips, or claustrophobia. Dual Energy Contrast Enhanced Digital Mammography (DE CEDM) is an investigational procedure that uses a non-standard contrast in a regular digital mammography exam that has been changed to give the needed dual energy and image. DE CEDM is not FDA approved. It is our hope that DE CEDM will also be able to detect unknown tumors because it will also detect new blood vessels. It is less expensive than MRI, could be more available to patients, and can be done on patients with pacemakers and clips. Claustrophobia will not be a problem. We plan to see if (DE CEDM) will help us better see the breast tumor and size of the breast tumor. We will also want to see if DE CEDM can detect additional unsuspected disease in the breast with the known tumor and in the other breast without a known tumor.

ELIGIBILITY:
Inclusion Criteria:

* Women with newly diagnosed unilateral breast cancer proven through core biopsy or FNA who are planned to have (preoperative) MRI within 30 days of DE CEDM to assess extent of disease/multifocality. (All women will have bilateral digital mammography as per standard of care.) The preoperative MRI will be based on the surgeon's recommendation.
* Both breasts are present.
* Women consenting to a bilateral DE CEDM examination.

Exclusion Criteria:

* Women under 21.
* Women who have already had a lumpectomy. (Index lesion has been removed and therefore, not evaluable for the purpose of this study.)
* Women undergoing neoadjuvant chemotherapy, hormone treatment, or radiation therapy.
* Known pregnancy.
* Women who have a contraindication to the intravenous use of iodinated or gadolinium-chelated contrast agent.
* Women with breast implants.
* Women with pacemakers.
* Women with aneurysm clips that don't allow for MRI.
* Women too claustrophobic to undergo MRI.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To estimate additional measures of accuracy of DE CEDM and MRI, such as the predictive values and ROC curves where applicable, for detecting multifocal or multicentric disease in the ipsilateral breast. | within 3 weeks of each other and within 30 days of surgery
  Every attempt will be made to perform all imaging exams All examinations will be completed within 30 days of scheduled surgery

SECONDARY OUTCOMES:
To compare the sensitivity and specificity of DE CEDM with that of breast MRI in the detection of disease in the contralateral breast. | within 3 weeks of each other and within 30 days of surgery
  Every attempt will be made to perform all imaging exams All examinations will be completed within 30 days of scheduled surgery
To estimate the interobserver variability of DE CEDM. | within 3 weeks of each other and within 30 days of surgery
  Every attempt will be made to perform all imaging exams All examinations will be completed within 30 days of scheduled surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Jochelson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org